CLINICAL TRIAL: NCT00227721
Title: Phase II Trial of Weekly Gemcitabine and Docetaxel Combination Therapy for Relapsed Ovarian or Peritoneal Cancer
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Relapsed or Refractory Ovarian Epithelial or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Morris (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Morris, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445432; P30CA022453 (NIH); WSU-C-2713
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel & Gemcitabine hydrochloride (Experimental): Docetaxel, 40 mg/m2, 30 min IV infusion on Days 1 and 8, of a 21 day cycle Gemcitabine hydrochloride, 800mg/m2 30 min IV infusion on Days1 and 8, of a 21 day cycle
  Interventions: Drug: Docetaxel; Drug: Gemcitabine hydrochloride

INTERVENTIONS:
Drug: Docetaxel — 40 mg/m2, 30 minute IV infusion, Days 1 and 8, Every 21 days
  Other Names: Taxotere®
Drug: Gemcitabine hydrochloride — 800mg/m2, 30 minute IV infusion, Days 1 and 8, every 21 days
  Other Names: Gemzar ®

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with relapsed or refractory ovarian epithelial or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with platinum-sensitive or -resistant relapsed or refractory ovarian epithelial or peritoneal cavity cancer treated with gemcitabine and docetaxel.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the time to treatment failure and progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior treatment with a platinum-containing regimen (platinum-resistant disease vs platinum-sensitive disease).

Patients receive gemcitabine IV over 30 minutes and docetaxel IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 3 additional courses beyond CR (≥ 6 total courses of treatment).

PROJECTED ACCRUAL: Approximately 36-62 patients (19-29 for stratum I [platinum-resistant disease] and 17-33 for stratum II [platinum-sensitive disease]) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or peritoneal cavity cancer
* Relapsed or refractory disease after prior first-line therapy with a platinum-containing regimen

  * Platinum-sensitive or -resistant disease

    * Platinum resistance is defined as relapsed or progressive disease within 6 months after completion of a platinum-containing regimen
* Measurable or evaluable disease

  * Evaluable disease is defined as CA 125 > 70 U/mL that has doubled from a baseline determination confirmed by ≥ 2 separate blood samples taken > 4 weeks apart OR other evidence demonstrating progressive disease after initial treatment regimen

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * AST or ALT normal AND alkaline phosphatase (AP) ≤ 5 times upper limit of normal (ULN)
  * AST or ALT ≤ 1.5 times ULN AND AP ≤ 2.5 times ULN
  * AST or ALT ≤ 5 times ULN AND AP normal

Renal

* Creatinine clearance > 30 mL/min
* Creatinine < 2.5 mg/dL

Cardiovascular

* No congestive heart failure
* No second or third degree heart block
* No myocardial infarction within the past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy > grade 1
* No other malignancy within the past 2 years except adequately treated skin cancer or carcinoma in situ of the cervix
* No history of severe hypersensitivity reaction to drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Prior paclitaxel allowed
* No more than 1 prior chemotherapy regimen

  * First-line platinum-based chemotherapy followed by consolidation therapy in the setting of a clinical and serologic complete response is considered 1 regimen
* No prior gemcitabine or docetaxel

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* More than 28 days since prior and no other concurrent investigational drugs for this cancer
* No other concurrent treatment or alternative therapy for this cancer

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2011-06 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Morris, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Northern Virginia Pelvic Surgery Assoc, Annandale, Virginia

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel & Gemcitabine Hydrochloride
Started | 30
Completed | 29
Not Completed | 1
Not completed — On study, but never treated. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel & Gemcitabine Hydrochloride
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 57.5 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to the Combination of Gemcitabine and Docetaxel in Patients With Platinum Sensitive and Resistant Epithelial Ovarian or Peritoneal Cancer.
Time Frame: Disease status by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) or Gynecological Cancer Intergroup (GCIG) CA-125 criteria was assessed every two cycles from enrollment up to progression, death, or five years (whichever occurred first).
Measure: Number (90% Confidence Interval); unit: percentage of participants with CR or PR
Arm/Group | Docetaxel & Gemcitabine Hydrochloride
Number analyzed (Participants) | 29
percentage of participants with CR or PR | 62 [47 to 75]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival estimated using Kaplan-Meier's product-limit method.
Time Frame: Every two cycles until disease progression or death, assessed up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Docetaxel & Gemcitabine Hydrochloride
Number analyzed (Participants) | 30
months | 7.2 [0.03 to 28.9]

ADVERSE EVENTS:
Time Frame: From enrollment up to progression, death, or five years (whichever occurred first).
Description: 30 patients were consented but one was never treated with any drug. Therefore, all AEs are from the 29 treated patients but the all-cause mortality is from all patients (intend to treat).
Arm/Group | Docetaxel & Gemcitabine Hydrochloride
All-Cause Mortality (participants affected / at risk) | 25/30
Serious Adverse Events (participants affected / at risk) | 14/29
Other Adverse Events (participants affected / at risk) | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel & Gemcitabine Hydrochloride (N=29)
Absolute neutrophil count (ANC) (Investigations) | 14 (14)
White Blood Count (WBC) (Investigations) | 10 (10)
Platelets (Investigations) | 7 (7)
Fatigue (General disorders) | 6 (6)
Hemoglobin (HGB) (Investigations) | 3 (3)
Pain (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Infection w/o Neutropenia (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Elevated Aspartate aminotransferase (AST) (Investigations) | 1 (1)
Elevated total bilirubin (Investigations) | 1 (1)
Abnormal magnesium (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fluid Retention Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Abnormal electrolytes (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel & Gemcitabine Hydrochloride (N=29)
Absolute neutrophil count (ANC) (Infections and infestations) | 9 (9)
WBC (Blood and lymphatic system disorders) | 15 (15)
Platelets (Blood and lymphatic system disorders) | 15 (15)
Fatigue (General disorders) | 21 (21)
Hemoglobin (HGB) (Investigations) | 24 (24)
Pain (General disorders) | 16 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 13 (13)
Elevated aspartate aminotransferase (AST) (Investigations) | 6 (6)
Elevated total bilirubin (hyperbilirubinemia) (Investigations) | 3 (3)
Abnormal magnesium (Metabolism and nutrition disorders) | 5 (5)
Bloating (Gastrointestinal disorders) | 2 (2)
Hemorrhage (Blood and lymphatic system disorders) | 4 (4)
Fever (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (13)
Elevated Alanine Aminotransferase (ALT) (Investigations) | 7 (7)
Elevated creatinine/bun (Investigations) | 5 (5)
Sensory Neuropathy (Nervous system disorders) | 18 (18)
Albumin (Investigations) | 2 (2)
Glucose (Metabolism and nutrition disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No